CLINICAL TRIAL: NCT01917045
Title: Different Lipid Soluble Opioids for Gynecologic Laparoscopic Surgery Postoperative Patient-controlled Analgesia --- a Double Blind Randomized Study
Brief Title: Different Lipid Soluble Opioids for Gynecologic Laparoscopic Surgery Postoperative Patient-controlled Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, ZhouYan, M.D, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LSOPCA-021
Record Dates: First submitted 2013-06-14; First posted 2013-08-06 (Estimated); Last update posted 2013-08-06 (Estimated); Status verified 2013-08

CONDITIONS: Post Operative Pain Management
Keywords: sufentanil; morphine; postoperative pain control; body fat percentage; gynecology laparoscopic surgery; lipid solubility
MeSH Terms: interventions — Sufentanil; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- low body fat percentage (Experimental): body fat percentage less than 30%
  Interventions: Drug: Sufentanil (R30730, brand name Sufenta); Drug: Sufentanil (R30730, brand name Sufenta) + Morphine; Drug: Morphine
- heigh body fat percentage (Experimental): body fat percentage more than 30%
  Interventions: Drug: Sufentanil (R30730, brand name Sufenta); Drug: Sufentanil (R30730, brand name Sufenta) + Morphine; Drug: Morphine

INTERVENTIONS:
Drug: Sufentanil (R30730, brand name Sufenta) — sufentanil 1ug/ml
Drug: Sufentanil (R30730, brand name Sufenta) + Morphine — sufentanil 0.5ug/ml+morphine 0.25mg/ml
Drug: Morphine — morphine 0. 5mg/ml

SUMMARY:
The investigators noticed that Body Fat Ratio might have great influence on the efficacy of different lipid soluble anesthetics. The objective of this clinical trial was to compare the effect of that Body Fat Ratio on the efficacy of different lipid soluble anesthetics.

DETAILED DESCRIPTION:
The objective of this clinical trial was to compare the effect of that Body Fat Ratio on the efficacy of different lipid soluble anesthetics.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists grade I-II
* adults aged over 20 and below 50 years old,
* non-smoker,
* with normal hepatic and renal function.

Exclusion Criteria:

* smoker ,
* any kind of mental disorder or
* history use of analgesics for more than 10 consecutive days,
* asthma; and
* those with digestion tract disorder who would get nausea or vomiting much more easily than normal people.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2012-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
visual analogue pain scores | 24hour
  we evaluate visual analogue pain scores at different time points within 24 hours after surgery

SECONDARY OUTCOMES:
nausea & vomiting | 24hour
  we evaluate nausea & vomiting at different time points within 24 hours after surgery. we ask the patient if she feel nausea or/and occured vomit, if so, 1 time will be recorded in the time point for incidence.

CONTACTS AND LOCATIONS:
Overall Officials: zhou yan, MD, Principal Investigator — PKU 1st hospital